CLINICAL TRIAL: NCT05353972
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of IMG-007 in Healthy Participants
Brief Title: Evaluate IMG-007 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inmagene LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMG-007-101
Record Dates: First submitted 2022-04-18; First posted 2022-04-29 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1 (Experimental): Single dose of IMG or placebo solution, intravenously administered
  Interventions: Drug: IMG-007 or placebo
- Cohort 2 (Experimental): Single dose of IMG or placebo solution, intravenously administered
  Interventions: Drug: IMG-007 or placebo
- Cohort 3 (Experimental): Single dose of IMG or placebo solution, intravenously administered
  Interventions: Drug: IMG-007 or placebo
- Cohort 4 (Experimental): Single dose of IMG or placebo solution, intravenously administered
  Interventions: Drug: IMG-007 or placebo
- Cohort 5 (Experimental): Single dose of IMG or placebo solution, intravenously administered
  Interventions: Drug: IMG-007 or placebo
- Cohort 6 (Experimental): Single dose of IMG or placebo solution, intravenously administered
  Interventions: Drug: IMG-007 or placebo
- Cohort 7 (Experimental): Single dose of IMG or placebo solution, intravenously administered
  Interventions: Drug: IMG-007 or placebo

INTERVENTIONS:
Drug: IMG-007 or placebo — intravenously administered

SUMMARY:
This first in human (FIH) study will evaluate the safety, tolerability, pharmacokinetics (PK)), and immunogenicity of a single ascending dose of IMG-007 in healthy participants.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled, sequential ascending, single dose escalating (SAD) study to assess the safety and PK profile of IMG-007 in healthy participants. The study is comprised of 3 phases: screening phase, treatment phase, and safety follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged between 18 to 50 years (inclusive)
2. Body mass index (BMI) greater than or equal to 18.0 kg/m2 and less than 32 kg/m2 and a minimum body weight of 50 kg for males and 45 kg for females at both the Screening and Baseline visits.
3. Able to participate and comply with all study procedures and restrictions, and willing to provide written informed consent to participate in the study.

Exclusion Criteria:

1. History of disease of the central nervous system, cardiovascular system, kidney, liver, digestive system, respiratory system, or metabolic/endocrine system
2. History of immunological abnormality
3. History of severe immediate hypersensitivity reaction to OX40 antagonists or other monoclonal antibodies
4. History of anaphylaxis or significant reactions to foods, medications, or other allergens
5. Major surgery ≤4 weeks before Baseline visit.
6. History of malignancy or known current malignancy,
7. Participant has an active infection or history of infections
8. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or antibody to Hepatitis B core antigen (HBcAb) with positive test for HBV DNA (>500 IU/ml) or hepatitis C antibodies (HCV) at Screening visit.
9. History of asthma
10. Having evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)
11. Participants with positive testing for COVID-19 at the Baseline visit.
12. Participants with clinically significantly abnormal laboratory values, as determined by the Investigator or medically qualified designee, i
13. Clinically significant abnormal findings at Screening or Baseline visits
14. Systolic blood pressure below 100 mmHg, at any time points prior to IMP administration
15. Use of any prescription medication
16. Use of over-the-counter medication
17. History of, or current substance abuse considered significant
18. Use of more than 5 tobacco/nicotine-containing products
19. Average alcohol consumption of more than 14 units/week for females and 21 units/week for males
20. Receipt of an investigational drug or medical device within 30 days or 5 half-lives (whichever is longer) prior to Day 1 dosing.
21. Live (attenuated) vaccination within 8 weeks before Screening or plan to be vaccinated by live (attenuated) vaccine during the trial
22. COVID-19 vaccination, or influenza vaccination(inactivated), within 14 days prior or planning to receive COVID-19 vaccination or influenza vaccination(inactivated) within 14 days post IMP administration.
23. Donated or lost more than 500 mL of blood or plasma within 3 months of Screening or received blood products within 8 weeks of Screening.
24. Pregnant or lactating women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | Cohort 1 to 5: up to 85 days; Cohort 6 to 7: up to 127 days;
  Incidence and severity of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) after infusion | Cohort 1 to 5: up to 85 days; Cohort 6 to 7: up to 127 days;
  Maximum observed concentration (Cmax) after infusion
Time at which Cmax is observed after infusion (tmax) | Cohort 1 to 5: up to 85 days; Cohort 6 to 7: up to 127 days;
  Time at which Cmax is observed after infusion (tmax)
Area under the concentration time curve from time 0 to last observation (AUC 0-t) | Cohort 1 to 5: up to 85 days; Cohort 6 to 7: up to 127 days;
  Area under the concentration time curve from time 0 to last observation (AUC 0-t)
Area under the concentration time curve from time 0 to infinity (AUC0-inf) | Cohort 1 to 5: up to 85 days; Cohort 6 to 7: up to 127 days;
  Area under the concentration time curve from time 0 to infinity (AUC0-inf)
Half-life t½ | Cohort 1 to 5: up to 85 days; Cohort 6 to 7: up to 127 days;
  Half-life t½
Incidence of anti-drug antibody (ADA) after infusion | Cohort 1 to 5: up to 85 days; Cohort 6 to 7: up to 127 days;
  Incidence of anti-drug antibody (ADA) after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schrader, Principal Investigator — Linear
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia